CLINICAL TRIAL: NCT07382492
Title: Clinical Effect of Swedish Massage Versus Adjuvant Yoga on Blood Glucose Level in Children With Type 1 Diabetes Mellitus
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Zaytoonah University of Jordan (Other)
Responsible Party: Principal Investigator, Mohamed Saied Zidan, Doctor, Al-Zaytoonah University of Jordan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Swedish massage yoga type 1 DM
Record Dates: First submitted 2026-01-27; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Type 1 Diabetes; Type 1 Diabetes Mellitus
Keywords: Swedish massage , Yoga , Type 1 diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diabetic children who received Swedish massage (Experimental): Twenty-five diabetic children who received Swedish massage in addition to routine nursing care of the unit for diabetes.
  Interventions: Procedure: Swedish massage in addition to routine nursing care of the unit for diabetes.
- Diabetic children who received children's yoga exercises (Experimental): Twenty-five diabetic children who received children's yoga exercises in addition to routine nursing care of the unit for diabetes.
  Interventions: Procedure: yoga exercises in addition to routine nursing care of the unit for diabetes.

INTERVENTIONS:
Procedure: Swedish massage in addition to routine nursing care of the unit for diabetes. — Swedish massage in addition to routine nursing care of the unit for diabetes.
  Arms: Diabetic children who received Swedish massage
Procedure: yoga exercises in addition to routine nursing care of the unit for diabetes. — yoga exercises in addition to routine nursing care of the unit for diabetes
  Arms: Diabetic children who received children's yoga exercises

SUMMARY:
Swedish massage (SM) and yoga are complementary non-pharmacological techniques that have recently been used in managing chronic disorders such as type 1 diabetes mellitus (T1DM). Both techniques play an important role in reducing stress, which contributes to lowering blood glucose levels in children with T1DM. Objective: To investigate the effect of Swedish massage versus children's yoga exercises on blood glucose levels of children with T1DM

DETAILED DESCRIPTION:
Swedish massage (SM) and yoga are complementary non-pharmacological techniques that have recently been used in managing chronic disorders such as type 1 diabetes mellitus (T1DM). Both techniques play an important role in reducing stress, which contributes to lowering blood glucose levels in children with T1DM. Objective: To investigate the effect of Swedish massage versus children's yoga exercises on blood glucose levels of children with T1DM

Progressive muscle relaxation (PMR) is one of the best effective non-pharmacological techniques, which decreases stress in children because it influences mental and physical conditions. It can be applied by making the muscles maximally strain, and then loosening it until the muscle is relaxed. It is repeated until children acquire complete relaxation (Casman & Nurhaeni, 2018).

Progressive muscle relaxation leads to regulation of autonomic nervous system activity that potentially contributes to medical management of T1DM through improving in glycosylated hemoglobin level (HbA1c) (Paschali et al., 2020). Swedish massage and Progressive muscle relaxation had an effective role in decreasing blood glucose level in children with T1DM, so that the pediatric nurse should apply and educate care giver about Swedish massage and PMR techniques (Ismaili et al., 2018)

ELIGIBILITY:
Inclusion Criteria:

* Diabetic children's age: 6 - 12 years.
* Children who live in Cairo only.
* Free from other medical disorders as cardiac, renal, or any other metabolic disorder

Exclusion Criteria:

* Diabetic children who can't understand the order
* Diabetic patient's who have medical disorders as cardiac,renal and other metabolic disorders

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2026-01-08 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Fasting blood glucose | 6 weeks
  measures sugar in your blood after an 8-12 hour fast (only water allowed), primarily to check for diabetes or prediabetes by showing your baseline sugar levels, with normal being under 100 mg/dL, prediabetes 100-125 mg/dL, and diabetes 126 mg/dL or higher on two separate tests,

SECONDARY OUTCOMES:
Random Blood sugar | 6 weeks
  measures blood sugar levels at any time, without fasting, to screen for diabetes, with normal for healthy adults generally under 140 mg/dL (7.8 mmol/L). Levels between 140-199 mg/dL suggest prediabetes, while 200 mg/dL or higher often indicates diabetes,
Glycosylated Hemoglobin (HbA1c). | 6 weeks
  a blood test measuring average blood sugar levels over the past 2-3 months by showing the percentage of sugar-coated hemoglobin in red blood cells,

CONTACTS AND LOCATIONS:
Locations (1):
- Outpatient Clinics of Universities and Private Medical Centers in Cairo, Cairo, Cairo Governorate, Egypt